CLINICAL TRIAL: NCT04465734
Title: A Randomized, Open-Label, Controlled, Multicenter, Phase III Clinical Study to Compare the Efficacy and Safety of HLX10 (Anti-PD-1 Antibody) in Combination With HLX04 (Anti-VEGF Antibody) Versus Sorafenib as the First-line Treatment in Patients With Locally Advanced or Metastatic Hepatocellular Carcinoma (HCC)
Brief Title: A Clinical Study to Compare the Efficacy and Safety of HLX10 in Combination With HLX04 Versus Sorafenib as the First-line Treatment in Patients With Locally Advanced or Metastatic HCC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial used sorafenib as a control drug. It's not suitable now(after the A+T has been approved).The sponsor terminated the trial.
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX10-009-HCC301
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Locally Advanced or Metastatic; Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (treatment group) (Experimental): HLX10 in combination with HLX04
  Interventions: Drug: HLX10; Drug: HLX04
- B (control group) (Sham Comparator): sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: HLX10 — HLX10 is an innovative monoclonal antibody targeting PD-1，developed by Shanghai Henlius Biotech, Inc.
  Arms: A (treatment group)
Drug: HLX04 — HLX04 is an recombinant anti-VEGF humanized monoclonal antibody ，developed by Shanghai Henlius Biotech, Inc.
  Other Names: HLX04 ( anti-VEGF antibody )
  Arms: A (treatment group)
Drug: Sorafenib — Sorafenib is a multi-target, multi-kinase inhibitor capable.The standard treatment of HCC.
  Arms: B (control group)

SUMMARY:
This study is a randomized, double-blind, multicenter, phase III clinical study to compare the efficacy and safety of HLX10 + HLX04 vs Sorafenibas as the First-line Treatment in Patients with Locally Advanced or Metastatic HCC

Eligible subjects in this study will be randomized to Arm A or Arm B at 2:1 ratio as follows:

Arm A (treatment group): HLX10 + HLX04 Arm B (control group): sorafenib Randomization is stratified by: region (Asia (excluding Japan) vs. others), HBV infection vs. HCV infection vs. no HBV or HCV infection, portal vein invasion or/and extrahepatic spread (with vs.without), and ECOG (0 vs. 1).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the clinical study;
2. Aged ≥ 18 years and ≤ 75 years;
3. Patients with histopathologically or cytologically diagnosed locally advanced or metastatic and/or unresectable HCC , or patients with clinically diagnosed HCC according to the diagnostic criteria of the American Association for the Study of Liver Diseases (AASLD);
4. Barcelona Clinic Liver Cancer (BCLC) Stage C; or BCLC Stage B patients who are not candidates for radical surgery and/or locoregional therapy.
5. Received no prior systemic HCC treatment (including chemotherapy, treatment with sorafenib, regorafenib, lenvatinib, or other small-molecule antiangiogenic agents);
6. At least one measurable lesion by the IRRC (central radiography) as per RECIST v1.1
7. Normal major organ functions as defined

Exclusion Criteria:

1. Patients with known hepatobiliary cell carcinoma, mixed cell carcinoma, or fibrolamellar cell carcinoma;
2. History of hepatic encephalopathy;
3. Patients with portal hypertension complicated with upper gastrointestinal hemorrhage, or esophageal/gastric fundal varices with the red color sign, or high hemorrhage risk investigated by the investigator within 6 months before the randomization. Subjects must receive endoscopic examinations to rule out high hemorrhage risk (e.g. red color sign and severe varices) before enrollment.
4. Patients with portal vein invasion at the main portal branch (Vp4), inferior vena cava involvement, or right cardiac involvement of HCC based on imaging examination. Patients with portal vein invasion at the main portal branch but with unobstructed blood flow in the bilateral or unilateral branch can be enrolled;
5. Central nervous system (CNS) or leptomeningeal metastases;
6. Positive for both HBV-DNA and HCV-RNA;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
tumor assessment | defined as a period from randomization to death of the subject for any reason (up to approximately 24 months)
  Overall survival (OS): defined as a period from randomization to death of the subject for any reason.
tumor assessment | Baseline until disease progression or death, whichever occurs first (up to approximately 12 months)
  Progression-free survival (PFS) (assessed by the independent radiology review committee [IRRC] based on Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics committee of zhongshan hospital affiliated to fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: No